CLINICAL TRIAL: NCT06630208
Title: Effectiveness of Myofascial Release in Patients With Chronic Post Sternotomy Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mayar Kamal Shehata Madian, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005235
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Chronic Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Myofascial Release Therapy; Breathing Exercises; Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release + Breathing exercises + Pharmacological treatment (Experimental): It will include 30 patients, who will receive myofascial release for 5 days, with breathing exercises in addition to pharmacological treatment.
  Interventions: Other: Myofascial release; Other: Breathing exercises; Drug: Pharmacological treatment
- Pharmacological treatment (Active Comparator): It will include 30 patients, who will receive pharmacological treatment only.
  Interventions: Drug: Pharmacological treatment

INTERVENTIONS:
Other: Myofascial release — The experimental group will undergo a 5-day consecutive myofascial release treatment, administered as Osteopathic Manipulative Treatment (OMT), with each session lasting a maximum of 15 minutes. The treatment will consist of three phases targeting the entire mediastinum: Thoracic Inlet (Indirect) Myofascial Release, Rib Raising with continued stretch of the paraspinal muscles to the L2 vertebral level, and Soft Tissue Cervical Paraspinal Muscle Stretch with Suboccipital Muscle Release. Participants will be positioned in a supine posture to enhance diaphragmatic excursion, with each session following a fixed, prearranged sequence of these techniques.
  Arms: Myofascial release + Breathing exercises + Pharmacological treatment
Other: Breathing exercises — Following the 3 phases of myofascial release, breathing exercises will be done for patients.
  Arms: Myofascial release + Breathing exercises + Pharmacological treatment
Drug: Pharmacological treatment — Patients will take pharmacological treatment prescribed by the cardiologist.

SUMMARY:
The main aim of this study is to investigate the effectiveness of Myofascial release in patients with chronic sternotomy pain.

DETAILED DESCRIPTION:
Post-sternotomy pain syndrome (PSPS) is a prevalent disorder affecting a substantial proportion of patients who have undergone sternotomy surgery, with incidence rates ranging from 10% to 40%. Several mechanisms have been proposed to be responsible for the development of PSPS; for example, intercostal neuralgia from scar-entrapped neuroma, brachial plexus injury, ribs or costal fractures with incomplete healing, sternal wound infections and even hypersensitivity reaction to sternal wire. chronic post sternotomy pain (CPSP) can compromise quality of life, affecting their sleep patterns and impairing their working ability.

During the first week after coronary artery bypass grafting (CABG) surgery, vital capacity (VC) decreases by 30-60% and even up to 1 year this remains reduced by 12%. Reduced VC has a negative effect on exercise tolerance (Vo2max) and therefore it is important to optimize pulmonary function after CABG surgery. The decreased thoracic mobility after CABG still presents 12 months after surgery. Thoracic mobility and vital capacity were affected more when the left internal thoracic artery (LITA)-retractor was used and reduced thoracic mobility is related to diminished pulmonary function.

New therapeutic-rehabilitative proposals have been tried in cardiac patients. After cardiac surgery, it was found that the responses of the cardiovascular, and respiratory systems get better after neuromuscular manual therapy. The strong correlation between manual therapy and its effects, suggests that a central control mechanism could be activated by manual therapy.

Using Myofascial release (MFR) techniques may be beneficial for patients post-CABG and off-pump coronary artery bypass grafting (OPCAB) surgery. The advantages of MFR techniques are gentleness and non-invasiveness. During therapy one works with fascia structures, thus, not influencing bone structures directly, These techniques are comfortable and safe, they may be applied in acute conditions.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Post-sternotomy pain (CPSP), defined as discomfort at the thorax after cardiac surgery, persisting for at least 2 months, and without apparent cause (I.e., such as infection or the underlying disease that motivated the surgery).
* Age between 55 to 65 years old.
* All patients will be under full medical supervision.
* Adherence to informed consent.
* Cardiac sternotomy intervention

Exclusion Criteria:

* Neuromuscular disorders.
* Any Active hemorrhage.
* The presence of an unstable cardiac, pulmonary or cerebral pathology.
* Poor cognition and mentality.
* Patients with active contagious skin conditions
* Any Cardiopulmonary problems (eg. Uncontrolled hypertension, Heart Failure, Arrhythmia)
* Patients with malignancy.
* Any acute viral infection.
* Patients with ascites or end-stage liver or kidney failure.
* Patients will participate in other physiotherapy programs rather than the prescribed protocol.
* Chest infection in last 3 months.
* Patients with musculoskeletal problems like any bone fracture
* Osteoporotic patients.
* Any recent open wound in the chest are.
* Hemodynamic instability.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 5 days
  Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
Upper chest expansion | 5 days
  It will be obtained by subtracting the inspiratory diameter from the expiratory diameter, according to the designated anatomical markers.
Lower chest expansion | 5 days
  It will be obtained by subtracting the inspiratory diameter from the expiratory diameter, according to the designated anatomical markers.
Pressure pain threshold | 5 days
  Pressure algometers are useful for quantifying the pressure pain thresholds of muscles. The pressure pain threshold of a patient is judged to be abnormal when the pressure pain threshold was lower than the normal value or if the pressure pain threshold of a certain site was lower than that of the opposite site by at least 2 kg/cm2, or if it was less than 3 kg/cm2.

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | 5 days
  It will be assessed by a spirometer before and after treatment. The patient will be asked to take a deep inspiration to expire forcefully and rapidly as much as possible through the mouthpiece.
Forced expiratory volume at one second (FEV1) | 5 days
  It will be assessed by a spirometer before and after treatment. The patient will be asked to take a deep inspiration to expire forcefully and rapidly as much as possible through the mouthpiece.
FEV1/FVC | 5 days
  The ratio between the forced expiratory volume at one second (FEV1) and forced vital capacity (FVC) will be calculated before and after treatment.
6-min walk test (6 MWT) | 5 days
  The total distance walked in meters will be measured.
Katz Index of Independence in Activities of Daily Living (ADL) | 5 days
  The Katz ADL index measures the self-care tasks which include bathing, dressing, toileting, transferring to and from a chair, maintaining continence and feeding. Answers are given in a dichotomous manner - yes or no for each task. The scores indicate the levels of functional impairments; total score of 6 - full function, 3 to 5 - moderate functional impairment, and 2 or less - severe functional impairment.
Pittsburgh Sleep Quality Index (PSQI) | 5 days
  The PSQI was designed to evaluate overall sleep quality in these clinical populations. Each of the questionnaire's 19 self-reported items belongs to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Arabic version of the 12-item short-form health survey (SF-12) | 5 days
  It will be used to assess the quality of life. The Arabic version of the SF-12 is a reliable, easy-to-use, and valid tool to measure health-related quality of life in the general population.
The Readiness for Return to Work (RRTW) | 5 days
  The Readiness for Return to Work (RRTW) model attempts to describe the intricate process of returning to work after a long-term sickness absence. The scale comprises 22 questions, which are divided into 13 questions for those who are not back to work yet, and 9 questions for those who are currently back at work.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Mahdi Ahmad, PhD, Study Chair — Cairo University
Locations (1):
- Cairo University, Giza, Egypt